CLINICAL TRIAL: NCT06140706
Title: Feasibility of a Video Telehealth Model to Evaluate Home Use of Transcutaneous Spinal Cord Stimulation for Enhanced Upper Limb Function
Brief Title: Feasibility of Home Based Transcutaneous Spinal Cord Stimulation for Persons With SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: ONWARD Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Beatrice Jenny Kiratli PhD, Research Health Scientist, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-68905
Record Dates: First submitted 2023-11-08; First posted 2023-11-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Tetraplegia
Keywords: paralysis; exercise; telemedicine; spinal cord stimulation; physical activity
MeSH Terms: conditions — Quadriplegia; Paralysis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tSCS plus home tele-video support (Experimental): Cervical transcutaneous spinal stimulation during home tele-video visits
  Interventions: Behavioral: transcutaneous Spinal Cord Stimulation (tSCS)

INTERVENTIONS:
Behavioral: transcutaneous Spinal Cord Stimulation (tSCS) — Neurostimulation for upper extremity training, delivered through video telehealth, 8 weeks of home use for (i) feasibility and (ii) potential functional improvement.

SUMMARY:
The proposed study will focus on the feasibility of and effectiveness to a home-based program for persons with chronic SCI focused on upper limb training augmented with a transcutaneous neurostimulator supported via a video telehealth platform.

DETAILED DESCRIPTION:
The overarching goal of this study is to train participants with tetraplegia and their companion to operate a non-invasive surface applied neurostimulation unit (ONWARD, ARCex) while performing a prescriptive functional task based upper extremity home program for 2 months. Participants will be supported with video-telehealth to assist with any difficulties that may arise and to progress their upper extremity home program. Evaluations will assess the feasibility of this video telehealth supported model as measured by the ease of use of the technology (QUEST 2.0, NASA-TLX) as well as participants ability to attend and complete all the training visits. Changes in upper extremity physical function will be measured using validated clinical tools (GRASSP, CUE-Q, DASH, COPM) as well as detailed evaluation of upper extremity muscle activation from surface EMG and strength measurements of pinch and grasp.

The primary outcome measure of this study is feasibility, and the secondary outcome measure is to capture changes in upper extremity performance.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran
2. Age 18-65
3. All gender, any ethnicity
4. Cervical Spinal Cord Injury C2-8
5. American Spinal Injury Association (ASIA) Impairment Scale (AIS) B, C or D
6. GRASSP-Prehension Score >10 or GRASSP Strength Score >30
7. Greater than 1 year post injury
8. Able to identify a companion to assist with neurostimulator setup in home environment.
9. Internet connection to support video telehealth connection
10. Willingness to travel to the VA Palo Alto Medical Center

Exclusion Criteria:

1. Cardiopulmonary disease or cardiac symptoms,
2. Autonomic dysreflexia that is uncontrolled or severe,
3. Implanted medical device(s),
4. Uncontrolled spasms that could limit participation in exercise training,
5. Skin breakdown or active pressure injury in areas of electrode placement.
6. Participants must not be engaged in any concurrent drug or device trial
7. Pregnant, are planning to become pregnant, or breastfeeding
8. The study is not deemed safe or appropriate in the opinion of the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
NASA-TLX (NASA Task Load Index) | At 8 weeks (after completion of home program)
  Measures subjective mental work load & physical effort
QUEST 2.0 (Quebec User Evaluation of Satisfaction with assistive Technology) | At 8 weeks (after completion of home program)
  Measures usability of device (eg, adjustability, comfort, safety and effectiveness)

SECONDARY OUTCOMES:
GRASSP (The Graded Redefined Assessment of Strength Sensibility and Prehension) | At entry (Baseline) and repeated at 8 weeks (after completion of home program)
  Measures upper limb sensation, strength, and prehension
CUE-Q (Capabilities of Upper Extremity Function) | At entry (Baseline) and repeated at 8 weeks (after completion of home program)
  Measures functional limitation and difficulty in performing upper limb activities
DASH (Disabilities of the Arm, Shoulder, and Hand) | At entry (Baseline) and repeated at 8 weeks (after completion of home program)
  Measures upper limb function during ADL tasks, work activities, recreational sports, and pain-related limitations
COPM (Canadian Occupational Performance Measure) | At entry (Baseline) and repeated at 8 weeks (after completion of home program)
  Measures performance & satisfaction of self-identified activities in self-care, productivity and leisure

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Kiratli, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No